CLINICAL TRIAL: NCT01481454
Title: Safety and Immunogenicity of a Quadrivalent Influenza Vaccine Administered Via the Intramuscular Route in Child/Adolescent and Adult Subjects
Brief Title: Study of a Quadrivalent Influenza Vaccine Administered Intramuscularly in Children/Adolescents and Adults
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sanofi Pasteur, a Sanofi Company (Industry)
Responsible Party: Sponsor
Organization: Sanofi (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: GQM04; U1111-1122-2719 (Other: WHO); 2011-005101-79 (EudraCT Number)
Record Dates: First submitted 2011-11-23; First posted 2011-11-29 (Estimated); Last update posted 2013-03-29 (Estimated); Status verified 2013-03

CONDITIONS: Influenza
Keywords: Influenza; Quadrivalent Inactivated Influenza Vaccine; Trivalent Inactivated Influenza Vaccine
MeSH Terms: conditions — Influenza, Human | interventions — Influenza Vaccines

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- Group 1: QIV Lot 1 (Experimental): Participants will receive the Quadrivalent Influenza Vaccine (QIV) from Lot 1.
  Interventions: Biological: Quadrivalent Influenza Vaccine (split virion, inactivated)
- Group 2: QIV Lot 2 (Experimental): Participants will receive the Quadrivalent Influenza Vaccine (QIV) from Lot 2.
  Interventions: Biological: Quadrivalent Influenza Vaccine (split virion, inactivated)
- Group 3: QIV Lot 3 (Experimental): Participants will receive the Quadrivalent Influenza Vaccine (QIV) from Lot 3.
  Interventions: Biological: Quadrivalent Influenza Vaccine (split virion, inactivated)
- Group 4: TIV (Active Comparator): Participants will receive the Trivalent Influenza Vaccine (TIV).
  Interventions: Biological: 2011 to 2012 Trivalent Influenza Vaccine

INTERVENTIONS:
Biological: Quadrivalent Influenza Vaccine (split virion, inactivated) — 0.5 mL, Intramuscular
  Arms: Group 1: QIV Lot 1
Biological: Quadrivalent Influenza Vaccine (split virion, inactivated) — 0.5 mL, Intramuscular
  Arms: Group 2: QIV Lot 2
Biological: Quadrivalent Influenza Vaccine (split virion, inactivated) — 0.5 mL, Intramuscular
  Arms: Group 3: QIV Lot 3
Biological: 2011 to 2012 Trivalent Influenza Vaccine — 0.5 mL, Intramuscular
  Arms: Group 4: TIV

SUMMARY:
The aim of the study is to assess the safety profile of a quadrivalent influenza vaccine (QIV) and to demonstrate that 3 different industrial lots of QIV induce an equivalent immune response in children/adolescents (9 to 17 years of age) and adults (18 to 60 years of age).

Primary Objective:

* To describe the safety profile (injection site reactions and systemic events) of each vaccine during the 21 days following vaccination, and serious adverse events (including adverse events of special interest) throughout the study in all adult and child/adolescent participants.

Secondary Objectives:

* To demonstrate that the 3 different industrial lots of quadrivalent influenza vaccine (QIV) induce an equivalent immune response at 21 days post-vaccination in both age groups (lot consistency)
* To describe the compliance of the immunogenicity of QIV to the European Medicines Agency Note for Guidance (NfG) (CPMP/BWP/214/96) in each age group.

DETAILED DESCRIPTION:
All participants will receive a single injection of their assigned vaccine during Visit 1. They will be followed up for safety and immunogenicity through Day 21 post-vaccination (Visit 2), and also monitored for safety for up to 6 months post-vaccination.

ELIGIBILITY:
Inclusion Criteria:

* Aged 9 to 11 years (children), 12 to 17 years (adolescents), or 18 to 60 years (adults) on the day of inclusion
* For child/adolescent subjects, informed consent form has been signed and dated by the parent(s) (and subject, if applicable by local regulations), or another legally acceptable representative (and independent witness, if required by local regulations), and the assent form has been signed and dated by the subject (if applicable by the local Ethics Committee or country regulations). For adult subjects, informed consent form has been signed and dated by the subject (and an independent witness, if required by local regulations).
* Subject/subject and parent/legally acceptable representative is/are able to attend all scheduled visits and to comply with all trial procedures
* Covered by health insurance, if required by local regulation.

Exclusion Criteria:

* Subject is pregnant, or lactating, or of childbearing potential (to be considered of non-childbearing potential, a female must be pre-menarche or post-menopausal for at least 1 year, surgically sterile, or using an effective method of contraception or abstinence from at least 4 weeks prior to vaccination and until at least 4 weeks after vaccination)
* Participation at the time of study enrollment or planned participation during the present trial period in another clinical trial investigating a vaccine, drug, medical device, or medical procedure
* Receipt of any vaccine in the 4 weeks preceding trial vaccination or planned receipt of any vaccine in the 3 weeks following trial vaccination
* Previous vaccination against influenza with the 2012 Southern Hemisphere formulation or the 2011-2012 Northern Hemisphere formulation in the previous 6 months with either the trial vaccine or another vaccine
* Receipt of immune globulins, blood or blood-derived products in the past 3 months
* Known or suspected congenital or acquired immunodeficiency; or receipt of immunosuppressive therapy, such as anti-cancer chemotherapy or radiation therapy, within the preceding 6 months; or long-term systemic corticosteroid therapy (prednisone or equivalent for more than 2 consecutive weeks within the past 3 months)
* Known systemic hypersensitivity to any of the vaccine components, or history of a life-threatening reaction to the vaccines used in the trial or to a vaccine containing any of the same substances
* Self-reported thrombocytopenia, contraindicating intramuscular vaccination based on investigator's judgment
* Bleeding disorder, or receipt of anticoagulants in the 3 weeks preceding inclusion, contraindicating intramuscular vaccination based on investigator's judgment
* Deprived of freedom by an administrative or court order, or in an emergency setting, or hospitalized involuntarily
* Current alcohol abuse or drug addiction (for adolescent and adult subjects)
* Chronic illness that, in the opinion of the investigator, is at a stage where it might interfere with trial conduct or completion
* Moderate or severe acute illness/infection (according to investigator judgment) on the day of vaccination or febrile illness (temperature ≥ 38.0°C). A prospective subject should not be included in the study until the condition has resolved or the febrile event has subsided
* Identified as an investigator or employee of the investigator or study center with direct involvement in the proposed study, or identified as an immediate family member (i.e., parent, spouse, natural, or adopted child) of the investigator or employee with direct involvement in the proposed study.

Ages: 9 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 1701 (Actual)
Dates: Start 2012-03; Primary Completion 2012-10 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Percentage of participants reporting solicited injection site reactions and solicited systemic reactions during the trial | Day 0 to 7 post-vaccination
  Solicited Injection Site Reactions: Pain, Erythema, Swelling, Induration, and Ecchymosis. Solicited Systemic Reactions: Fever (Temperature), Headache, Malaise, Myalgia, and Shivering
Percentage of participants reporting unsolicited systemic reactions including serious adverse events (SAE) throughout the trial. | Day 0 up to six months post-vaccination
  An SAE is defined as any untoward medical occurrence that at any dose (including overdose): Results in death; Is life-threatening; Requires inpatient hospitalization or prolongation of existing hospitalization; Results in persistent or significant disability / incapacity; Is a congenital anomaly / birth defect; Is an important medical event.

SECONDARY OUTCOMES:
Percentage of participants with seroprotection and seroconversion post vaccination with either the investigational QIV, or TIV or the licensed 2011-2012 TIV | Day 21 post-vaccination
  Immunogenicity assessed by hemagglutination inhibition (HAI) assay for each vaccine strain.
  Seroprotection defined as a post-vaccination titer of ≥ 40 (1/dil); Seroconversion defined for participants with a pre-vaccination titer < 10 (1/dil) and a post-vaccination titer of ≥ 40 (1/dil).
Level of anti-hemagglutinin antibody titers for each of the 4 strains for each lot of the investigational QIV vaccine. | 21 Days post-vaccination

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Sanofi Pasteur SA
Locations (6):
- Australia (2):
  - Melbourne
  - Westmead NSW
- Philippines (4):
  - Calamba Laguna City
  - City of Muntinlupa
  - Malate, Manila
  - Quezon City

REFERENCES:
- [Derived] Cadorna-Carlos JB, Nolan T, Borja-Tabora CF, Santos J, Montalban MC, de Looze FJ, Eizenberg P, Hall S, Dupuy M, Hutagalung Y, Pepin S, Saville M. Safety, immunogenicity, and lot-to-lot consistency of a quadrivalent inactivated influenza vaccine in children, adolescents, and adults: A randomized, controlled, phase III trial. Vaccine. 2015 May 15;33(21):2485-92. doi: 10.1016/j.vaccine.2015.03.065. Epub 2015 Apr 2. PMID 25843270
- See also: Related Info — http://www.sanofipasteur.com